CLINICAL TRIAL: NCT04660058
Title: Associations Among Serum and Gastric Juice Bile Acid Profile, Bile Acid-microbiota Cross-talk in Stomach and the Development of Gastric Cancer: A Case-control Study
Brief Title: Associations Among Serum and Gastric Juice Bile Acid Profile, Bile Acid-microbiota Cross-talk in Stomach and the Development of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20202100-F-1
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bile Reflux; Gastric Cancer; Precancerous Lesion
Keywords: bile acid; gastric microbiota; Gastric Cancer; precancerous lesion
MeSH Terms: conditions — Bile Reflux; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — serum and gastric juice samples will not be retained; pathological tissue samples will be retained in Xijing Hospital
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic gastritis: patients with chronic non-atrophic gastritis and chronic atrophic gastritis according to histopathological results
- precancerous lesion: patients with gastric intestinal metaplasia and intraepithelial neoplasia according to histopathological results
- gastric cancer: patients with gastric cancer according to histopathological results

SUMMARY:
To explore the associations among bile acid profile, bile acid-microbiota cross-talk and the development of gastric cancer, so as to better prevent the occurrence and development of gastric cancer

DETAILED DESCRIPTION:
This study is a case-control study. Patients, according to the pathological results, will be consecutively enrolled and divided into gastric cancer group, gastric precancerous lesions group, and chronic gastritis group. The serum and gastric juice bile acid profiles, gastric microbial composition of each group patients will be detected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, gender is not limited;
2. No history of antibiotic or probiotic use for 8 weeks;
3. No preoperative chemotherapy or radiation therapy prior to the examination;
4. Voluntary intravenous blood collection, gastroscopy, extraction of gastric juice and pathological biopsy.
5. Voluntary testing for H. pylori

Exclusion Criteria:

1. had undergone upper gastrointestinal and colon surgery;
2. Previous diagnosis of Malignant Tumors;
3. Presence of a disease or medication that affects bile acid metabolism, such as endocrine or autoimmune diseases;
4. Recent use of drugs that affect gastrointestinal motility;
5. Presence of contraindications to endoscopy;
6. pregnant and lactating women;
7. Those with mental disorders;
8. Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients are from Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
corelation between the bile acid profile and gastric mucosa diseases | up to 6 months
  Investigators evaluate the corelation between the bile acid profile and gastric mucosa diseases according to the results of UPLC-MS/MS and pathological .
corelation between the bile acid profile and gastric microbiota in different groups | up to 6 months
  Investigators explore the cross-talk between bile acid and gastric microbiota according to the results of 16s rRNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China